CLINICAL TRIAL: NCT02195908
Title: The Comparative Study on the Effectiveness of Single Acupoint and Matching Acupoints.
Brief Title: The Different Effectiveness of Single Acupoint（PC6 or CV12) vs Matching Acupoints(PC6 and CV12) in Chemotherapy-induced Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: National Basic Research Program, China (Other)
Responsible Party: Principal Investigator, Yi Guo, the Dean of Acupuncture and Moxibustion College, Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CB543201-01
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: to Evaluate the Effectiveness of Acupucnture in the Management of Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Single point PC6 (Experimental): choose single point: Neiguan(PC6).Neiguan(PC6): On the anterior aspect of the forearm,between the tendons of the palmaris longus and the flexor carpi radialis, 2 B-cun proximal to the palmar wrist crease.Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA. The operation lasts for 30 min. The treatment is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  Interventions: Other: single point Neiguan(PC6) plus antiemetic drug
- Single point CV12 (Experimental): choose another single point Zhongwan（CV12）. Zhongwan(CV12): On the upper abdomen, 4 B-cun superior to the centre of the umbilicus, on the anterior median line. Manipulating until achieving a "de Qi" sensation, then the needle is connected through a electro-acupuncture apparatus,the positive pole is linked to the needle, and the reference pole is located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA.The operation lasts for 30 min. The treatment is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  Interventions: Other: single point Zhongwan(CV12) plus antiemetic drug
- Matching points PC6+CV12 (Experimental): Choose both Neiguan point(PC6) and Zhongwan point(CV12). Manipulating until achieving a "de Qi" sensation, then the needles are connected through a electro-acupuncture apparatus, the positive poles are linked to the needle, and the reference poles are located near the acupoint about 1cm with a paster. Frequency 10Hz,the intensity of stimulation is adjusted according to the patient's tolerance, and the electric current is less than 10mA. The operation lasts for 30 min. The treatment is scheduled to occur within 30min-60min before chemotherapy infusion for 4 days.
  Interventions: Other: matching points Neiguan(PC6) and Zhongwan(CV12) plus antiemetic drug
- only antiemetic (Active Comparator): The control group will receive standard antiemetic alone. Standard antiemetic for all groups is based on American Society of Clinical Oncology clinical practice guideline. 5-hydroxytryptamine-3 (5-HT3) antagonist (Ramosetron, Tropisetron) and dexamethasone are supplied from the first day of chemotherapy, and lasting for 3-5 days.
  Interventions: Drug: only antiemetic drug

INTERVENTIONS:
Other: single point Neiguan(PC6) plus antiemetic drug
  Arms: Single point PC6
Other: single point Zhongwan(CV12) plus antiemetic drug
  Arms: Single point CV12
Other: matching points Neiguan(PC6) and Zhongwan(CV12) plus antiemetic drug
  Arms: Matching points PC6+CV12
Drug: only antiemetic drug
  Arms: only antiemetic

SUMMARY:
The purpose of this study is to clarify whether the matching acupoints are more effective than a single point by electro-acupuncture in the management of chemotherapy-induced nausea and vomiting .

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed as cancer and need to accept chemotherapy.
2. The score of Karnofsky ≥70
3. Patients of either gender and older than 18 years
4. Patients receiving chemotherapy both outpatients and inpatients
5. Patients receiving chemotherapy either the first or multiple cycle, but the patient will be taken in only one time
6. To receive chemotherapy containing cisplatin(DDP≥75mg/m2) or joint chemotherapy programmes of Anthracyclines(Adriamycin≥40mg/m2 or epirubicin≥60mg/m2)
7. Life expectancy≥ 6 months
8. Willing to participate in the study and be randomized into one of the four study groups.

Exclusion Criteria:

1. To receive radiotherapy and chemotherapy
2. Gastrointestinal tumors
3. Patients with serious liver disease or abnormal hepatorenal function (AST,ACT, and TBIL are 3 times more than normal, BUN and Cr are 2 times more than normal)
4. Presence of cardiac pacemaker
5. Active skin infection
6. Nausea and/or vomiting resulting from opioids or metabolic imbalance (electrolyte disturbances)
7. Patients unable to provide self-care or communication
8. Nausea and/or vomiting resulting from mechanical risk factors (i.e., intestinal obstruction)
9. Brain metastases
10. Women in pregnant and lactating period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the frequency of Nausea and Vomiting | 6days

SECONDARY OUTCOMES:
the grading of constipation and diarrhea | 3 weeks
electrogastrogram | 3 weeks
the assessment of quality of life | 3 weeks
the assessment of Anxiety and Depression | 3 weeks

OTHER OUTCOMES:
blood routine examination | 3 weeks
electrocardiogram | 3 weeks
hepatic and renal function | 3 weeks
other adverse effect during the chemotherapy | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of TCM, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Chen B, Hu SX, Liu BH, Zhao TY, Li B, Liu Y, Li MY, Pan XF, Guo YM, Chen ZL, Guo Y. Efficacy and safety of electroacupuncture with different acupoints for chemotherapy-induced nausea and vomiting: study protocol for a randomized controlled trial. Trials. 2015 May 12;16:212. doi: 10.1186/s13063-015-0734-x. PMID 25963295